CLINICAL TRIAL: NCT02354872
Title: Optimized Chronic Care for Smokers: A Comparative Effectiveness Approach; Motivation Project: Testing Intervention Components for the Smoker Who is Unwilling to Quit
Brief Title: Motivation Project: Testing Intervention Components for the Smoker Who is Unwilling to Quit
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Penn State University (Other); University of Illinois at Chicago (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 2014-1041Motivation; A534252 (Other: UW Madison); SMPH\MEDICINE\TOBACCO RE (Other: UW Madison); 1P01CA180945-01 (NIH); CTRI (Other: UW Madison)
Record Dates: First submitted 2015-01-22; First posted 2015-02-03 (Estimated); Last update posted 2020-09-22 (Actual); Status verified 2020-09

CONDITIONS: Smoking; Motivation; Smoking Cessation
Keywords: Nicotine
MeSH Terms: conditions — Smoking; Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (16):
- Mini-Lozenge, BR, 5Rs, BA (Experimental): 1; This arm of the project will address the following question: How effective is the following intervention? Mini-Lozenge, BR, 5Rs, BA
  Interventions: Drug: Nicotine Mini-Lozenge; Behavioral: Behavioral Reduction Counseling; Behavioral: 5Rs Motivation Counseling; Behavioral: Behavioral Activation Counseling
- Mini-Lozenge, BR, 5Rs, No BA (Experimental): 2; This arm of the project will address the following question: How effective is the following intervention? Mini-Lozenge, BR, 5Rs, No BA
  Interventions: Drug: Nicotine Mini-Lozenge; Behavioral: Behavioral Reduction Counseling; Behavioral: 5Rs Motivation Counseling
- Mini-Lozenge, BR, No 5Rs, BA (Experimental): 3; This arm of the project will address the following question: How effective is the following intervention? Mini-Lozenge, BR, No 5Rs, BA
  Interventions: Drug: Nicotine Mini-Lozenge; Behavioral: Behavioral Reduction Counseling; Behavioral: Behavioral Activation Counseling
- Mini-Lozenge, BR, No 5Rs, No BA (Experimental): 4; This arm of the project will address the following question: How effective is the following intervention? Mini-Lozenge, BR, No 5Rs, No BA
  Interventions: Drug: Nicotine Mini-Lozenge; Behavioral: Behavioral Reduction Counseling
- Mini-Lozenge, No BR, 5Rs, BA (Experimental): 5; This arm of the project will address the following question: How effective is the following intervention? Mini-Lozenge, No BR, 5Rs, BA
  Interventions: Drug: Nicotine Mini-Lozenge; Behavioral: 5Rs Motivation Counseling; Behavioral: Behavioral Activation Counseling
- Mini-Lozenge, No BR, 5Rs, No BA (Experimental): 6; This arm of the project will address the following question: How effective is the following intervention? Mini-Lozenge, No BR, 5Rs, No BA
  Interventions: Drug: Nicotine Mini-Lozenge; Behavioral: 5Rs Motivation Counseling
- Mini-Lozenge, No BR, No 5Rs, BA (Experimental): 7; This arm of the project will address the following question: How effective is the following intervention? Mini-Lozenge, No BR, No 5Rs, BA
  Interventions: Drug: Nicotine Mini-Lozenge; Behavioral: Behavioral Activation Counseling
- Mini-Lozenge, No BR, No 5Rs, No BA (Experimental): 8; This arm of the project will address the following question: How effective is the following intervention? Mini-Lozenge, No BR, No 5Rs, No BA
  Interventions: Drug: Nicotine Mini-Lozenge
- No Mini-Lozenge, BR, 5Rs, BA (Experimental): 9; This arm of the project will address the following question: How effective is the following intervention? No Mini-Lozenge, BR, 5Rs, BA
  Interventions: Behavioral: Behavioral Reduction Counseling; Behavioral: 5Rs Motivation Counseling; Behavioral: Behavioral Activation Counseling
- No Mini-Lozenge, BR, 5Rs, No BA (Experimental): 10; This arm of the project will address the following question: How effective is the following intervention? No Mini-Lozenge, BR, 5Rs, No BA
  Interventions: Behavioral: Behavioral Reduction Counseling; Behavioral: 5Rs Motivation Counseling
- No Mini-Lozenge, BR, No 5Rs, BA (Experimental): 11; This arm of the project will address the following question: How effective is the following intervention? No Mini-Lozenge, BR, No 5Rs, BA
  Interventions: Behavioral: Behavioral Reduction Counseling; Behavioral: Behavioral Activation Counseling
- No Mini-Lozenge, BR, No 5Rs, No BA (Experimental): 12; This arm of the project will address the following question: How effective is the following intervention? No Mini-Lozenge, BR, No 5Rs, No BA
  Interventions: Behavioral: Behavioral Reduction Counseling
- No Mini-Lozenge, No BR, 5Rs, BA (Experimental): 13; This arm of the project will address the following question: How effective is the following intervention? No Mini-Lozenge, No BR, 5Rs, BA
  Interventions: Behavioral: 5Rs Motivation Counseling; Behavioral: Behavioral Activation Counseling
- No Mini-Lozenge, No BR, 5Rs, No BA (Experimental): 14; This arm of the project will address the following question: How effective is the following intervention? No Mini-Lozenge, No BR, 5Rs, No BA
  Interventions: Behavioral: 5Rs Motivation Counseling
- No Mini-Lozenge, No BR, No 5Rs, BA (Experimental): 15; This arm of the project will address the following question: How effective is the following intervention? No Mini-Lozenge, No BR, No 5Rs, BA
  Interventions: Behavioral: Behavioral Activation Counseling
- No Mini-Lozenge, No BR, No 5Rs, No BA (Experimental): 16; This arm of the project will address the following question: How effective is the following intervention? No Mini-Lozenge, No BR, No 5Rs, No BA
  Interventions: Other: No Treatment

INTERVENTIONS:
Drug: Nicotine Mini-Lozenge — If randomized to only the Nicotine Mini-Lozenge condition: Participants randomized to this condition will receive up to a 12 month supply of 2 mg or 4 mg nicotine mini-lozenges. Mini-Lozenges will be given at the initial visit and over the course of the whole study. Participants will be instructed to use 9 pieces daily for the 12 months.
  Arms: Mini-Lozenge, BR, 5Rs, BA; Mini-Lozenge, BR, 5Rs, No BA; Mini-Lozenge, BR, No 5Rs, BA; Mini-Lozenge, BR, No 5Rs, No BA; Mini-Lozenge, No BR, 5Rs, BA; Mini-Lozenge, No BR, 5Rs, No BA; Mini-Lozenge, No BR, No 5Rs, BA; Mini-Lozenge, No BR, No 5Rs, No BA
Behavioral: Behavioral Reduction Counseling — We will deliver BR in 10 (10-15 minute) sessions over a 52-week period, with an in-person session at Visit 1 followed by nine phone counseling sessions. Sessions are front-loaded to enhance acquisition of new behaviors. BR Counseling will emphasize the development of smoking control skills via feasible, specific, and graded assignments of smoking reduction activities that will be tracked over time. BR will also emphasize competence and self-efficacy, both which will be directly linked to the practice of smoking reduction skills and success in smoking control. The health counselor will provide rationales for the reduction intervention, why reduction (e.g., eliminating smoking contexts) should help the smoker, and provide the participant with specific exercises and goals. The health counselor will explicitly address pragmatic issues such as work contexts, smoking policies, and habits that interfere with smoking reduction efforts.
  Arms: Mini-Lozenge, BR, 5Rs, BA; Mini-Lozenge, BR, 5Rs, No BA; Mini-Lozenge, BR, No 5Rs, BA; Mini-Lozenge, BR, No 5Rs, No BA; No Mini-Lozenge, BR, 5Rs, BA; No Mini-Lozenge, BR, 5Rs, No BA; No Mini-Lozenge, BR, No 5Rs, BA; No Mini-Lozenge, BR, No 5Rs, No BA
Behavioral: 5Rs Motivation Counseling — The 5Rs Motivation Counseling will be delivered in four (10-15 min) sessions over a 52-week period. Participants in the "on" condition will receive three brief phone sessions over the year to prompt processing of motives for smoking reduction or cessation. The health counselor and smoker will discuss: 1) Relevance of smoking to the individual; 2) Risks of continued heavy smoking; 3) Rewards of quitting and significant reduction; and 4) Roadblocks to success; and will do so on a 5) Repeated basis. The discussion will follow the general principles of MI: counselors will use strategies that are nonauthoritarian, nonconfrontational, supportive, and use open-ended questions.
  Arms: Mini-Lozenge, BR, 5Rs, BA; Mini-Lozenge, BR, 5Rs, No BA; Mini-Lozenge, No BR, 5Rs, BA; Mini-Lozenge, No BR, 5Rs, No BA; No Mini-Lozenge, BR, 5Rs, BA; No Mini-Lozenge, BR, 5Rs, No BA; No Mini-Lozenge, No BR, 5Rs, BA; No Mini-Lozenge, No BR, 5Rs, No BA
Behavioral: Behavioral Activation Counseling — The BA treatment will be delivered in 10 (10-15 minute) sessions over a 52-week period starting with Visit 1 followed by nine phone counseling sessions. This BA treatment will be modeled after Behavioral Activation for quitting smoking, but made relevant for smoking reduction. Treatment goals focus on helping participants engage in positively reinforcing activities while not smoking. The treatment includes: 1) a rationale for the BA exercises as they relate to smoking (e.g., engaging in non-smoking reinforcers will provide other sources of pleasure and assist with cutting down); 2) assessment of the participant's goals, values, and reinforcing value of current nonsmoking activities; 3) training in self-monitoring using an activity log; 4) ongoing assignments of activities that should significantly increase the participant's nonsmoking reinforcement and create broader lifestyle and cue exposure changes; and 5) problem-solving to address obstacles to goal attainment.
  Arms: Mini-Lozenge, BR, 5Rs, BA; Mini-Lozenge, BR, No 5Rs, BA; Mini-Lozenge, No BR, 5Rs, BA; Mini-Lozenge, No BR, No 5Rs, BA; No Mini-Lozenge, BR, 5Rs, BA; No Mini-Lozenge, BR, No 5Rs, BA; No Mini-Lozenge, No BR, 5Rs, BA; No Mini-Lozenge, No BR, No 5Rs, BA
Other: No Treatment — No Treatment
  Arms: No Mini-Lozenge, No BR, No 5Rs, No BA

SUMMARY:
The ultimate goal of this research is to develop a chronic care treatment package for smokers that will address the challenges and opportunities of each phase of the cessation process - motivation, preparation, cessation, maintenance, and relapse recovery. That is, to develop treatments for smokers not yet ready to quit, those who are preparing to quit, those actively engaged in the quitting process and those who have tried to quit but relapsed. To achieve this goal, this research comprises three distinct research studies, each of which represent a phase in a comprehensive chronic care treatment model for clinical intervention with smokers in the primary care setting: the Motivation Study, the Cessation Study, and the Long-term Quitting Study. The goal of each study is to test and identify effective intervention components for distinct phases of the smoking cessation process. These components will then be combined for future research on the effectiveness of this chronic care treatment package. This study is a 2x2x2x2 factorial design. Participants will be randomized to one of two levels on four different factors: 1) Nicotine Mini-Lozenge vs. No Mini-Lozenge, 2) Behavioral Reduction Counseling (intervention: BR) vs. No Behavioral Reduction Counseling, 3) 5Rs Motivation Counseling (intervention 5 R's) vs. No 5Rs Motivation Counseling, and 4) Behavioral Activation Counseling (intervention BA) vs. No Behavioral Activation Counseling. These components have strong theoretical and empirical support, but their relative, additive, and interactive effects are unknown.

ELIGIBILITY:
Inclusion Criteria:

* age >=18 years; smoking >4 cigarettes/day for the previous 6 months; able to read, write, and speak English; have reliable phone access and agree to respond to Interactive Voice Response (IVR) phone prompts; and if currently using NRT, agreeing to use only study medication for the duration of the study. We will not exclude participants based on their prior use of cessation medication or if they use multiple tobacco products in order to enhance real-world generalization (these will be statistically controlled in analyses); not currently attempting to quit smoking; not intending to quit smoking (defined as no plans to quit in the next month); and planning to remain in the intervention catchment area for at least 12 months.

Exclusion Criteria:

* currently taking bupropion or varenicline; medical contraindications to using NRT including hospitalized (for at least one night) for a stroke, heart attack, congestive heart failure or diabetes in the last 30 days; diagnosis of or treatment for schizophrenia, a psychotic disorder or bipolar disorder in the last 10 years; and, if the participant is a woman of childbearing potential, being pregnant or intending to becoming pregnant or unwillingness to use an approved method of birth control during treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 577 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2019-03-19 (Actual); Study Completion 2019-03-19 (Actual)

PRIMARY OUTCOMES:
7-Day Point-Prevalence Abstinence | 12 months
  Participants who self-report no smoking for the past 7 days at the assessment endpoint (12 month follow-up) will be considered to meet criteria for 7-Day Point-Prevalence Abstinence. Participants who who report any smoking in the past 7 days (at the 12 month follow-up) will be considered to be relapsed (smoking).

CONTACTS AND LOCATIONS:
Overall Officials: Michael C Fiore, MD, MPH, MBA, Study Chair — University of Wisconsin Center for Tobacco Research and Intervention, School of Medicine and Public Health; Jessica Cook, PhD, Study Director — University of Wisconsin Center for Tobacco Research and Intervention, School of Medicine and Public Health; Robin Mermelstein, PhD, Principal Investigator — Institute for Health Research and Policy, University of Illinois at Chicago
Locations (1):
- University of Wisconsin Center for Tobacco Research and Intervention, School of Medicine and Public Health, Madison, Wisconsin, United States

REFERENCES:
- [Derived] Cook JW, Baker TB, Fiore MC, Collins LM, Piper ME, Schlam TR, Bolt DM, Smith SS, Zwaga D, Jorenby DE, Mermelstein R. Evaluating four motivation-phase intervention components for use with primary care patients unwilling to quit smoking: a randomized factorial experiment. Addiction. 2021 Nov;116(11):3167-3179. doi: 10.1111/add.15528. Epub 2021 May 19. PMID 33908665
- See also: University of Wisconsin Center for Tobacco Research and Intervention, School of Medicine and Public Health — http://www.ctri.wisc.edu/